CLINICAL TRIAL: NCT03637907
Title: Spectral Computed Tomography With Photon Counting Detector of Brain and Vessels.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Staffan Holmin, Professor, Karolinska Institutet
Other Study IDs: KI-KTH-20180111
Record Dates: First submitted 2018-03-16; First posted 2018-08-20 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Tomography; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not applicable - no intervention. — No intervention is performed, just a CT with a new detector and comparison with the same patients older image.

SUMMARY:
Primary purpose of the study is to show wether computed tomography with photon counting detector has a diagnostic image quality as good as, or better than classic computed tomography in investigations concerning stroke work-up.

DETAILED DESCRIPTION:
Images of the skull/brain at the level of the inner ear/temporal bone and the level of nucleus lentiformis will be compared with the same patients routine brain done in TIA (transient ischemic attack)/stroke workup.

Images of the carotid plaque will be compared with the same patients routine CT-angiogram done in TIA/stroke workup.

ELIGIBILITY:
Inclusion Criteria:

* Brain exam with CT and/or CT neck/brain vessels prior to this study. Regarding neck-vessel imaging - carotid stenosis of 30% or more. Normal kidney function.

Exclusion Criteria:

* no contraindications to iodine contrast for neck-vessel imaging with contrast.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in the ordinary stroke workup that do both CT brain and CTA of neck/brain vessel will be asked if we can ask them to participate in this study. Of the ones with carotid stenosis 30% or more we will ask patients to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2018-01-11 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Equal or better images vs classic computed tomography. | During 2020
  Are images taken with photon counting detector of brain and vessels worse, equal or better in comparison with ordinary computed tomography.
  Comparison of images with kernals (or algorithms) for bone and soft tissue at the level of the carotid plaque, inner ear/hindbrain and nucl lentiformis.
  Comparison of the ability of the spectral function - the ability to separate iodine, soft tissue and calcifications- if applicable.
  The comparison will be done as a grading (better, equal or worse) regarding the different kernals compared to routine CT exams from the same patient.
  Significance of difference between proportions with thh use of Fisher's exact test or Pearson's χ2 as appropriate. Evaluation with Cohen´s kappa with 95% CI to assess the level of inter-reader agreement

SECONDARY OUTCOMES:
Diagnostic information in comparison with MRI | During 2020
  If MRI are performed of the patients brain and/or vessels - a comparison how the diagnostic information is/are relative images from MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed, contact the Principal Investigator for (anonymous) data